CLINICAL TRIAL: NCT00387972
Title: A Multi-center, Double-blind, Parallel-group, Randomized, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Denagliptin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study Of Denagliptin In Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study cancelled before enrollment
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPB107246
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus (T2DM); glycosylated hemoglobin (HbA1c); denagliptin; diabetes treatment; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — denagliptin

INTERVENTIONS:
Drug: denagliptin (GW823093)

SUMMARY:
GW823093 is a selective DPP-IV Inhibitor and is being investigated as a once a day oral therapy. The purpose of the Study is to evaluate the effectiveness, safety, and tolerability of 2 doses of GW823093, compared to placebo, taken once daily in patients with Type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus treated with diet and exercise or oral anti-diabetic treatment
* Body mass index between 20 and 40
* Females of childbearing potential must use adequate birth control.

Exclusion criteria:

* Subjects with previous use of insulin
* Type 1 diabetes
* Uncontrolled thyroid disease
* History of drug or alcohol abuse in the past year
* Any other clinically significant disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2007-10 (Estimated); Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in blood glucose regulation after 26 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in glycemic parameters, insulin, body weight and waist circumference, and safety measures

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, DM, FRCP, Study Director — GlaxoSmithKline
Locations (55):
- United States (55):
  - GSK Clinical Trials Call Center, Tallassee, Alabama
  - GSK Clinical Trials Call Center, Phoenix, Arizona
  - GSK Clinical Trials Call Center, Tucson, Arizona
  - GSK Clinical Trials Call Center, Beverly Hills, California
  - GSK Clinical Trials Call Center, Carmichael, California
  - GSK Clinical Trials Call Center, Concord, California
  - GSK Clinical Trials Call Center, Torrance, California
  - GSK Clinical Trials Call Center, Victorville, California
  - GSK Clinical Trials Call Center, Wilmington, Delaware
  - GSK Clinical Trials Call Center, Boynton Beach, Florida
  - GSK Clinical Trials Call Center, Clearwater, Florida
  - GSK Clinical Trials Call Center, Coral Gables, Florida
  - GSK Clinical Trials Call Center, Hialeah, Florida
  - GSK Clinical Trials Call Center, Hollywood, Florida
  - GSK Clinical Trials Call Center, Melbourne, Florida
  - GSK Clinical Trials Call Center, Miami, Florida
  - GSK Clinical Trials Call Center, Opa-locka, Florida
  - GSK Clinical Trials Call Center, Plantation, Florida
  - GSK Clinical Trials Call Center, Tampa, Florida
  - GSK Clinical Trials Call Center, Calhoun, Georgia
  - GSK Clinical Trials Call Center, Roswell, Georgia
  - GSK Clinical Trials Call Center, Hayden Lake, Idaho
  - GSK Clinical Trials Call Center, Chicago, Illinois
  - GSK Clinical Trials Call Center, Lake Zurich, Illinois
  - GSK Clinical Trials Call Center, Watseka, Illinois
  - GSK Clinical Trials Call Center, Baton Rouge, Louisiana
  - GSK Clinical Trials Call Center, Marrero, Louisiana
  - GSK Clinical Trials Call Center, Oxon Hill, Maryland
  - GSK Clinical Trials Call Center, Detroit, Michigan
  - GSK Clinical Trials Call Center, City of Saint Peters, Missouri
  - GSK Clinical Trials Call Center, Florissant, Missouri
  - GSK Clinical Trials Call Center, St Louis, Missouri
  - GSK Clinical Trials Call Center, Las Vegas, Nevada
  - GSK Clinical Trials Call Center, Williamsville, New York
  - GSK Clinical Trials Call Center, Charlotte, North Carolina
  - GSK Clinical Trials Call Center, Morehead City, North Carolina
  - GSK Clinical Trials Call Center, Fargo, North Dakota
  - GSK Clinical Trials Call Center, Cincinnati, Ohio
  - GSK Clinical Trials Call Center, Columbus, Ohio
  - GSK Clinical Trials Call Center, Guthrie, Oklahoma
  - GSK Clinical Trials Call Center, Norman, Oklahoma
  - GSK Clinical Trials Call Center, Oklahoma City, Oklahoma
  - GSK Clinical Trials Call Center, Yukon, Oklahoma
  - GSK Clinical Trials Call Center, Eugene, Oregon
  - GSK Clinical Trials Call Center, Medford, Oregon
  - GSK Clinical Trials Call Center, Beaver Falls, Pennsylvania
  - GSK Clinical Trials Call Center, Fleetwood, Pennsylvania
  - GSK Clinical Trials Call Center, Warminster, Pennsylvania
  - GSK Clinical Trials Call Center, Anderson, South Carolina
  - GSK Clinical Trials Call Center, Chattanooga, Tennessee
  - GSK Clinical Trials Call Center, Johnson City, Tennessee
  - GSK Clinical Trials Call Center, Cleburne, Texas
  - GSK Clinical Trials Call Center, San Antonio, Texas
  - GSK Clinical Trials Call Center, Seguin, Texas
  - GSK Clinical Trials Call Center, Weber City, Virginia